CLINICAL TRIAL: NCT00823654
Title: Multi-Center Study of Serum Biomarkers to Characterize the Effects of Therapy on Ovarian Reserve in Premenopausal Women With Early-stage Breast Cancer BRCA Mutations
Brief Title: Serum Biomarkers to Characterize the Effects of Therapy on Ovarian Reserve in Premenopausal Women With Early-stage Breast Cancer or BRCA Mutations
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Yale University (Other); New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-156
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer
Keywords: Breast; Questionaires; Blood draw; BRCA1; BRCA2; 08-156
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood

GROUPS / COHORTS (2):
- Premenopausal Women with Early Stage Breast Cancer
  Interventions: Other: Blood draw and questionnaires
- Unaffected High Risk Women with BRCA mutations
  Interventions: Other: Blood draw and questionnaires

INTERVENTIONS:
Other: Blood draw and questionnaires — Identify eligible premenopausal patients and obtain informed consent ↓ Register patients at Memorial Sloan Kettering Cancer Center
  ↓ Baseline evaluation: Blood draw and baseline reproductive health questionnaire (Appendix A)/menstrual calendar (Appendix C) / sexual health questionnaires (Appendices E, F, G)
  ↓ Start planned therapy (or observation)
  ↓ Evaluation at completion of chemotherapy Blood draw and collection of monthly menstrual calendars
  ↓ One year post chemo Blood draw and collection of monthly menstrual calendars/follow-up reproductive health questionnaire (Appendix B)
  ↓ Annual follow-up x 3 years Blood draw and collection of monthly menstrual calendars/follow-up reproductive health questionnaire (Appendix B) )/ sexual health questionnaires (Appendices E, F, G)
  Groups: Premenopausal Women with Early Stage Breast Cancer
Other: Blood draw and questionnaires — Identify eligible premenopausal patients and obtain informed consent ↓ Register patients at Memorial Sloan Kettering Cancer Center
  ↓ Baseline evaluation: Blood draw and baseline reproductive and sexual health questionnaires (Appendices A, E, F, G)/menstrual calendar (Appendix C)
  ↓ Year 1 follow up Blood draw and collection of monthly menstrual calendars (Appendix C)/follow-up reproductive and sexual health questionnaires (Appendices B, E, F, G)
  ↓ Annual follow-up years x 3 if feasible Blood draw and collection of monthly menstrual calendars (Appendix C)/follow-up reproductive and sexual health questionnaires (Appendices B, E, F, G)
  Groups: Unaffected High Risk Women with BRCA mutations

SUMMARY:
The purpose of this study is to learn more about the effects of your BRCA mutation on the ovaries. The BRCA gene can make it hard to conceive a child in the future. It may also bring on early menopause. The researchers will check blood levels of hormones that the ovaries produce. The hormones that researchers will check are anti-Mullerian hormone (AMH), estradiol and follicle stimulating hormone (FSH). The researchers will do this before, during, and after cancer treatment. The researchers will also ask you to fill out questionnaires about your menstrual cycle (your periods) and information about your health and pregnancies. This may help us learn which women will be more likely to have early menopause.

ELIGIBILITY:
Inclusion Criteria:

For Premenopausal Women with Early Stage Breast Cancer

1. Participant is between 18-44 years old.
2. Participant is premenopausal.
3. Participant is female.
4. Participant has a known breast cancer diagnosis of AJCC Stage 0-III breast cancer, regardless of hormone-receptor status or HER2-overexpression, before the start of planned adjuvant or neoadjuvant chemotherapy and/or hormonal therapy.
5. The chemotherapy regimen must be either CMF, anthracycline-containing, or taxane-containing. If hormonal therapy is planned, the regimen must be limited to tamoxifen All biologics are allowed in addition to the above therapies.
6. The participant has regular menstrual cycles; note: patients can have no more than 1 irregular cycle (too early or too late) within the past year and/or at least 10 spontaneous cycles within the past year. Exceptions are made for patients who have been pregnant in the last 12 months and patients with IUDs or a LARC.

Subject Inclusion:

For Unaffected High Risk Premenopausal Women with BRCA mutations

1. The participant is between 25 and 45 years of age.
2. The participant is female.
3. The patient has a known BRCA mutation.
4. Have regular menstrual (21-35 days); patients can have no more than 1 irregular cycle (too early or too late) within the past year or were pregnant in the past 12 months, and/or at least 10 spontaneous cycles within the past year. Exceptions are made for patients who have been pregnant in the last 12 months and patients with IUDs or a LARC.

Subject Inclusion:

For affected BRCA1 and BRCA2 mutation carriers, affected women with non-BRCA mutations, and BC patients with no mutations (control)

1 . Premenopausal women age 21-45 with stage 0-3 breast cancer. 2. No prior ovarian surgery or ovarian disease. 3. No prior chemotherapy. 4. Regular menstrual periods (21-35 days), no PCOS. 5. No hormonal contraception within the prior 4 weeks. 6. Mutation testing decision based on NCCN Guidelines V1.2021: according to these Guidelines, both centers test all pre-menopausal women with breast cancer for BRCA and non-BRCA mutations which are the subject of this proposal.

7. Receiving an anthracycline (typically doxorubicin/Adriamycin) and Cy (AC)-based chemotherapy protocol.

Exclusion Criteria:

For Cohort of Premenopausal Women with Early Stage Breast Cancer

* Prior therapy for breast cancer or any other cancer, such as chemotherapy, hormonal therapy or immunotherapy.
* Ovarian resection, unilateral or bilateral oophorectomy, hysterectomy or radiation to pelvic region.
* Plans for risk-reducing bilateral oophorectomy within one year of completion of chemotherapy.
* Prior known infertility; infertility is defined as one year of inability to conceive despite unprotected intercourse and/or the need to use medication (e.g clomiphene) or assisted reproductive technology (e.g. intrauterine insemination or in vitro fertilization) to attempt pregnancy.
* Family history of a first-degree relative with non-surgical menopause < age 40
* Current pregnancy.

Subject Exclusion Criteria:

For Unaffected High Risk Premenopausal Women with BRCA mutation

1. Participant has therapy for breast cancer or any other cancer, such as chemotherapy, hormonal therapy or immunotherapy.
2. Participant has ovarian resection, unilateral or bilateral oophorectomy, radiation to pelvic region.
3. Participant has Plans for risk-reducing bilateral oophorectomy within one year of completion of chemotherapy.
4. Participant has prior known infertility; infertility is defined as one year of inability to conceive despite unprotected intercourse and/or the need to use medication (e.g., clomiphene) or assisted reproductive technology (e.g., intrauterine insemination or in vitro fertilization) to attempt pregnancy.
5. Participant has a family history of a first-degree relative with non-surgical menopause < age 40.
6. Participant is currently pregnant. For affected BRCA1 and BRCA2 mutation carriers, affected women with non-BRCA mutations, and BC patients with no mutations (control)

1. Subjects who did not undergo mutation testing, as well as those who tested positive for more than one family (BRCA1, BRCA2, non-BRCA) of ATM-Pathway gene mutations, will be excluded.

2. Women aged >42 years will be excluded as they carry a very high probability of chemotherapy-induced OI49. It is important to select an age range where immediate OI is less likely to occur because if most women become menopausal post-chemotherapy, the comparison of ovarian reserve decline will not be feasible. 3. In our prior grant period, we showed that the AC-based and CMF regimens similarly compromise ovarian reserve (Fig. 1)9 Currently, the AC-based chemotherapy is utilized in >90% breast ca cases, and CMF protocol is rarely administered9. For this reason and to enhance uniformity, rare non-AC-based protocols will be excluded. 4. A previous study showed that smoking and BRCA mutations may have additive negative effects on the age of menopause27, consequently, we will exclude current smokers (smoked 100 cigarettes lifetime and currently smokes, per CDC). Based on our past studies6,9, the smoking incidence is low in our study population (<20%) and should not significantly limit accrual.

5. BMI: In our recent publication9 (Fig. 1), the mean BMI was 24.22 ±0.4 (median 23.2; range 17-42); hence the extreme BMI values are rare in our population. Nevertheless, those with BMI of <18.5 and >40 will be excluded.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of premenopausal women with early-stage breast cancer will be recruited from the Breast Cancer Service at MSKCC and New York Presbyterian Hospital-Weill Medical College of Cornell University. In addition, breast cancer patients seeking consultation with a reproductive endocrinologist to address issues of fertility preservation prior to the start of therapy will be offered participation (Dr. Oktay at Yale Medicine.
  Patients of unaffected high risk premenopausal women with BRCA mutations will be recruited from the Breast Cancer Services especially the high risk surveillance clinics at MSKCC and New York Presbyterian Hospital-Weill Medical College of Cornell Univeristy.
Sampling Method: Non-Probability Sample
Enrollment: 609 (Estimated)
Dates: Start 2009-01 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
characterize the changes in serum AMH from baseline to 1 year post-chemo (or 1 year into hormonal therapy if no chemotherapy planned) | 2 years
  in premenopausal breast cancer patients & to characterize the changes in serum AMH from baseline to 1 year in unaffected high risk BRCA mutation carriers.

SECONDARY OUTCOMES:
To characterize the changes in serum estradiol and FSH from baseline to one year postchemotherapy (or 1 year into hormonal therapy if no chemotherapy planned) in premenopausal breast cancer patients and BRCA mutation carriers. | 2 years
To characterize the changes over time in serum AMH, estradiol, and FSH in premenopausal breast cancer patients and unaffected high risk BRCA mutation carriers. | 2 years
To describe the impact of commonly used therapies for early-stage breast cancer on self-reported monthly menstrual cycles and future pregnancy/reproductive health. | 2 years
To study the differences in ovarian reserve between BRCA1+ and BRCA2+ women. | 2 years
To study sexual health and function in unaffected high risk BRCA mutation carriers | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari Goldfarb, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Oktay KH, Bedoschi G, Goldfarb SB, Taylan E, Titus S, Palomaki GE, Cigler T, Robson M, Dickler MN. Increased chemotherapy-induced ovarian reserve loss in women with germline BRCA mutations due to oocyte deoxyribonucleic acid double strand break repair deficiency. Fertil Steril. 2020 Jun;113(6):1251-1260.e1. doi: 10.1016/j.fertnstert.2020.01.033. Epub 2020 Apr 22. PMID 32331767
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org